CLINICAL TRIAL: NCT06498804
Title: The Blood Patch in the Management of Intracranial Hypotension: Description of a Population and Professional Practices
Brief Title: The Blood Patch in the Management of Intracranial Hypotension
Acronym: BPIH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9059
Record Dates: First submitted 2024-04-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Intracranial Hypotension
Keywords: Intracranial Hypotension; post-dural puncture headache; cranial nerve symptoms; hearing disturbances; vertigo
MeSH Terms: conditions — Intracranial Hypotension; Post-Dural Puncture Headache; Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intracranial hypotension results from leakage and/or hypotension of cerebrospinal fluid. It can be spontaneous or secondary to a dural puncture complicating perimedullary anesthesia or a lumbar puncture. The incidence remains low with less than 1% post spinal puncture (25 gauge needle), but is observed more frequently following a lumbar puncture, up to 36% with a 20 or 22 gauge needle. Accidental puncture of the dura mater with a 17 gauge needle used for epidural anesthesia is associated with postpuncture headaches in 75-80% of cases. Classically, symptoms appear 24 to 48 hours after the puncture and consist of very intense, postural, fronto-occipital headaches which may be associated with cranial nerve symptoms such as visual or hearing disturbances or vertigo. Among the risk factors are the size and type of the needle, age under 60 and female gender. About 90% of PDPH are self-limiting within 7-10 days.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject having benefited from a bloodpatch between 01/01/2021 and 12/31/2022

Exclusion Criteria:

- Subject (and/or their legal representative if applicable) having expressed their (their) opposition to the reuse of their data for scientific research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) having benefited from a bloodpatch between 01/01/2021 and 12/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Descriptions of professional practices in the management of intracranial hypotension by blood patch at the University Hospitals of Strasbourg | Through study completion, an average of 2 months
  This retrospective study focuses on the description of the practices of doctors at the Strasbourg University Hospital in the management of intracranial hypotension by blood patch.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation médecine Péri-Opératoire - CHU de Strasbourg - France, Strasbourg, France